CLINICAL TRIAL: NCT00336219
Title: COMPETITION: Investigation of Clinical Endpoints for Treatment-induced Gastroesophageal Reflux Disease (GERD) Symptom Changes
Brief Title: Symptom Assessment in Adult Patients With Erosive GERD (Gastroesophageal Reflux Disease) or enGERD (Endoscopic-negative GERD) After Treatment With Pantoprazole (BY1023/M3-343)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/M3-343
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-10

CONDITIONS: GERD
Keywords: GERD; Pantoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

ARMS (1):
- 1 (Active Comparator): Pantoprazole 40 mg
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Symptom Assessment after treatment with Pantoprozole 40 mg

SUMMARY:
The aim of this study is to compare investigator and patient-assessed gastroesophageal reflux disease symptoms in patients with erosive GERD or endoscopic-negative GERD (enGERD). An endoscopy will be performed at study start and study end. During the study, the patients will complete a patient-orientated, self-assessed reflux questionnaire (ReQuest™ questionnaire). The study duration consists of a baseline period (8 days) and treatment period (28 days). Pantoprazole (tablet) will be administered once daily at one dose level. The study will provide further data on safety and tolerability of pantoprazole.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Outpatients
* History of GERD-related symptoms for at least 6 months prior to study inclusion
* Endoscopically confirmed erosive GERD or non-erosive GERD

Main Exclusion Criteria:

* Acute peptic ulcer and/or ulcer complications
* PPIs during last 7 days prior to study start
* Systemic glucocorticoids or non-steroidal anti-inflammatory drugs including COX-2 inhibitors during the last 28 days prior to study start; except regular intake of acetylsalicylic acid up to a daily dose of 163 mg/day
* Intake of PPIs in combination with antibiotics for eradication of H. pylori

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
symptom assessment as measured by ReQuest™ questionnaire and investigator. | 28 days

SECONDARY OUTCOMES:
symptom assessment on days 7, 14, and 28 as measured by ReQuest™ questionnaire and investigator | 28 days
endoscopic healing after 28 days | 28 days
health-related quality of life after 28 days | 28 days
safety. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Holtmann, Prof., Principal Investigator — Department of Gastroenterology, Hepatology and General Medicine, Royal Adelaide Hospital, North Terrace, Adelaide, Australia
Locations (37):
- Australia (4):
  - Altana Pharma/Nycomed, Bondi Junction
  - Altana Pharma/Nycomed, Box Hill, Victoria
  - Altana Pharma/Nycomed, New South Wales
  - Altana Pharma/Nycomed, South Australia
- Austria (5):
  - Altana Pharma/Nycomed, Feldbach
  - Altana Pharma/Nycomed, Graz
  - Altana Pharma/Nycomed, Stockerau
  - Altana Pharma/Nycomed, Vienna
  - Altana Pharma/Nycomed, Wiener Neustadt
- Germany (20):
  - Altana Pharma/Nycomed, Amberg
  - Altana Pharma/Nycomed, Aschersleben
  - Altana Pharma/Nycomed, Berlin
  - Altana Pharma/Nycomed, Cologne
  - Altana Pharma/Nycomed, Freising
  - Altana Pharma/Nycomed, Germersheim
  - Altana Pharma/Nycomed, Grünstadt
  - Altana Pharma/Nycomed, Jülich
  - Altana Pharma/Nycomed, Köthen
  - Altana Pharma/Nycomed, Künzing
  - Altana Pharma/Nycomed, Landsberg
  - Altana Pharma/Nycomed, Langen
  - Altana Pharma/Nycomed, Leipzig
  - Altana Pharma/Nycomed, Ludwigshafen
  - Altana Pharma/Nycomed, Lüneburg
  - Altana Pharma/Nycomed, Mönchengladbach
  - Altana Pharma/Nycomed, München
  - Altana Pharma/Nycomed, Potsdam-Babelsberg
  - Altana Pharma/Nycomed, Reinfeld
  - Altana Pharma/Nycomed, Saarbrücken
- Hungary (8):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Győr
  - Altana Pharma/Nycomed, Hatvan
  - Altana Pharma/Nycomed, Kaposvár
  - Altana Pharma/Nycomed, Kistarcsa
  - Altana Pharma/Nycomed, Miskolc
  - Altana Pharma/Nycomed, Szentes
  - Altana Pharma/Nycomed, Vác